CLINICAL TRIAL: NCT02077660
Title: The Effect of Green Tea on Anthropometric, Oxidation and Inflammation Parameters in Physically Active Elderly Compared to Sedentary Elderly
Brief Title: Green Tea Effect on Anthropometric, Oxidation and Inflammation Parameters in Physically Active vs. Sedentary Elders
Acronym: GT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 01; Rambam MC (Other: Rambam MC)
Record Dates: First submitted 2014-02-12; First posted 2014-03-04 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Aging
Keywords: Green tea, aging, oxidation, anthropometrics.

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 daily placebo tea bags for 12 weeks (Placebo Comparator): All subjects will undergo a 12 weeks supplemented with four daily placebo maltodextrin "tea-bags". The subjects will be instructed than to brew the placebo sachets for five minute in 240 mL boiling water without stirring and to drink 4 cups per day for 12 weeks period (Placebo period).
  Interventions: Other: 4 daily placebo tea bags for 12 weeks
- Four green tea bags per day for 12 weeks (Experimental): After the placebo period, all subjects will undergo a 12 weeks supplemented with four daily green tea bags. The subjects will be instructed than to brew the green tea sachets for five minute in 240 mL boiling water without stirring and to drink 4 cups per day for 12 weeks period (Green tea period).
  Interventions: Dietary Supplement: Four green tea bags per day for 12 weeks

INTERVENTIONS:
Dietary Supplement: Four green tea bags per day for 12 weeks — Four green tea bags per day for 12 weeks
  Arms: Four green tea bags per day for 12 weeks
Other: 4 daily placebo tea bags for 12 weeks — 4 daily placebo tea bags for 12 weeks
  Arms: 4 daily placebo tea bags for 12 weeks

SUMMARY:
The purpose of this study is to evaluate the beneficial effects of a long term (12 weeks) green tea drinking on plasma, erythrocytes and saliva oxidative stress biomarkers and antioxidant capacity, as well as on cardiometabolic risk factors: anthropometric, inflammation and metabolic parameters in a healthy aging men and women.

DETAILED DESCRIPTION:
A prospective, crossover trial in which every individual served its own control. All subjects undergo a four weeks washout period, during which they briefed to avoid tea drinking and antioxidant supplements until the end of the study. At the end of the washout period, blood and saliva samples is collected after 12 hours of night fast. Subsequently, all subjects receive the maltodextrin containing placebo "tea bags". The subjects instructed to brew the placebo sachets for five minute in 240 mL boiling water without stirring and to drink 4 cups per day for 12 weeks period (placebo period). After the placebo period, fasting samples collected once more and the subjects receive the green tea bags. Preparation and drinking instructions are the same as the placebo drink. At the end of the 12 weeks, green tea drinking, fasting blood and saliva samples drawn for the third time. During the study, every 4 weeks the subjects get additional placebo or green tea bags. Assessment of nutritional consumption of macronutrients and antioxidants using a food diary, physical activity lifestyle as well as weight, body fat and circumference measurements is made at the beginning, middle and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Age: 60-76 Years
* Able to understand the meaning of Informed Consent procedure and willing to consent

Exclusion Criteria:

* Any active disease state
* Unstable chronic disease (diabetes, vascular, renal)

Ages: 60 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Plasma protein carbonyls | 24 weeks
  Protein carbonyls, nmol/mg
Plasma thiobarbituric acid reactive substance | 24 weeks
  Thiobarbituric acid reactive substance , nmol/mL
Plasma lipid peroxides | 24 weeks
  Lipid peroxides, nmol/mL
Erythrocytes catalase | 24 weeks
  Catalase activity, milliunits/mg
Erythrocytes resistance to oxidative hemolysis | 24 weeks
  hemolysis test, percentage
Saliva enzymatic antioxidants | 24 weeks
  Oral peroxidase activity, milliunits/mg
Saliva antioxidant capacity | 24 weeks
  Total antioxidant capacity, millimolar/mg

SECONDARY OUTCOMES:
Total body weight | 24 weeks
  Body weight, kg
Total body fat percentage | 24 weeks
  Body fat, %
Body circumference | 24 weeks
  Waist and hip circumference, cm
Serum inflammatory status | 24 weeks
  Serum C-reactive protein mg/dL
Saliva inflammatory status Saliva matrix metalloproteinase 8 (MMP8) | 24 weeks
  Saliva matrix metalloproteinase 8, µg/L
Saliva inflammatory status - saliva interleukin 8 (IL8) | 24 weeks
  Saliva interleukin 8, ng/L

CONTACTS AND LOCATIONS:
Overall Officials: Yishai Levy, Professor, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam MC, Haifa, Israel